CLINICAL TRIAL: NCT05561608
Title: Validation of Heart Rate Recovery as a Peri-operative Risk Measure (VERVE)
Brief Title: Validation of Heart Rate Recovery as a Peri-operative Risk Measure
Acronym: VERVE
Status: Completed | Type: Observational
Sponsor: University of Glasgow (Other)
Collaborators: NHS National Waiting Times Centre Board (Other); NHS Greater Glasgow and Clyde (Other); NHS Ayrshire and Arran (Other); NHS Lanarkshire (Other Government)
Responsible Party: Principal Investigator, Dr Ben Shelley, Honorary Clinical Associate Professor/Consultant in Cardiothoracic Anaesthesia and Intensive Care, University of Glasgow
Other Study IDs: 21/WA/0207
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Peri-operative Injury
Keywords: Heart rate recovery; Submaximal exercise testing; Post-operative myocardial injury; Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Is heart rate recovery after submaximal exercise (i.e. not to exhaustion) a valid risk measure for post-operative outcomes?

DETAILED DESCRIPTION:
There are approximately 1.5 million major operations carried out in the NHS every year. As the population ages, and surgical technique becomes more advanced, more patients are undergoing operations which carry a high risk of complications. Currently, doctors predict this risk by asking patients about medical problems and their level of physical fitness. If an operation is very high risk, a patient may undergo cardiopulmonary exercise testing (CPET) where the patient rides an exercise bike to maximum effort (exhaustion) whilst their heart and lung function is measured. This gives the doctor specific numbers which can be discussed with the patient about the risk of complications after surgery. However, CPET is expensive and not all patients are able to do it, for example due to joint or circulation problems. Patients can also find attempting to reach maximal effort demanding and uncomfortable.

Heart rate recovery (HRR) after maximal exercise has been shown to indicate post-operative risk of complications, and is also related to life-expectancy in people with heart failure. The utility of HRR after submaximal exercise however has not been investigated as extensively. One group demonstrated that submaximal HRR predicts post-operative complications after lung surgery, and submaximal HRR also predicts life-expectancy in healthy individuals. There is less information about submaximal HRR as the methods of measuring it are not standardised. Previous work by our group has confirmed the reproducibility of submaximal HRR in a healthy population, and demonstrated different ways in which to measure it. The investigators believe that submaximal HRR provides a "middle-ground" method of assessing how fit a patient is for surgery.

With informed consent, 95 patients across four hospitals in the West of Scotland will perform a step test pre-operatively. The step test will involve non-invasive measurement of the heart rate. Patients will exercise until approximately two-thirds of their predicted maximum heart rate is reached and then recover sitting, whilst the rate of their heart rate recovery is recorded. Patients will have pre- and post-operative troponin values measured (blood marker of strain/injury to the heart). Alongside the blood tests, patients will also answer questionnaires related to their quality of life, and information regarding other post-operative complications will be recorded.

The study aims to demonstrate that submaximal HRR is predictive of post-operative myocardial injury (stress/injury to the heart wall due to the body's response to the operation) and that is it a valid measure when compared to the scores, blood tests and exercise tests that are currently in use in the NHS. In the future, submaximal exercise testing with HRR measurement may be offered to patients unable to perform CPET and will guide shared decision-making between patient, surgeon and anaesthetist to ensure the best outcome for the patient regarding their surgical options.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Age 50 years or over
* Able to walk unaided
* Planned elective intermediate/high risk surgery as defined by the ESC/ESA guidelines (i.e. >1% risk of mortality)

Exclusion Criteria:

* Pregnancy
* Ongoing participation in any investigational research which could undermine the scientific basis of the study
* Presence of any of the American Thoracic Society's contraindications to exercise testing
* Previous intermediate/high risk surgery within three months prior to recruitment
* Previous participation in the VERVE study at any time

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 95 patients 50 years or over undergoing intermediate/high risk surgery in the West of Scotland. Patients will be recruited from the Golden Jubilee National Hospital, Queen Elizabeth University Hospital, University Hospital Hairmyres or University Hospital Crosshouse.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Post-operative myocardial injury | 48 hours post-operatively
  Post-operative troponin over the 99th centile upper reference limit plus a 20% change (increase or decrease)

SECONDARY OUTCOMES:
Acute Kidney Injury | 1 week post-operatively
  As defined by KDIGO consensus
Major adverse kidney events | 30 days post-operatively
  Composite of renal mortality, renal replacement therapy, over 30% decline in eGFR from baseline
Cardiovascular complications | 7 days post-operatively
  Incidence of myocardial infarction, cardiac death, non-fatal cardiac arrest, coronary revascularisation, pulmonary embolus, deep-veined thrombosis, or new onset atrial fibrillation
Major adverse cardiac events | 30 days post-operatively
  Composite of cardiac death, myocardial infarction, non-fatal cardiac arrest, and coronary revascularisation
Infective complications | 7 days post-operatively
  Presence of fever <38.5 and clinical suspicion of infection
Neurological complications | 7 days post-operatively
  Delirium or stroke
Pulmonary complications | 7 days post-operatively
  Atelectasis, pneumonia, acute respiratory distress syndrome or pulmonary aspiration
Quality of recovery scale - 15 | 2 days post-operatively
EQ-5D-5L | 30 days and 1 year post-operatively
  Patient reported quality of life score
Days alive and out of hospital | 30 days post-operatively
Length of hospital stay (with/without hospital mortality) | Up to 1 year post-operatively
Readmission to hospital | Within 30 days post-operatively
Admission/re-admission to Intensive Care | 14 days post-operatively
Mortality | Day 30, day 90 and 1 year post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Shelley, MBChB, MD, Principal Investigator — National Waiting Times Centre Board
Locations (3):
- United Kingdom (3):
  - Golden Jubilee National Hospital, Clydebank
  - University Hospital Hairmyres, East Kilbride
  - University Hospital, Crosshouse, Kilmarnock

IPD SHARING:
Plan to Share IPD: Yes
We are keen to provide opportunities for data sharing. All requests for data sharing will be assessed individually and requests complying with the data governance regulations of the Sponsor and NHS R&D will be honoured.
Supporting Information: Study Protocol, SAP, Analytic Code

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT05561608/Prot_SAP_000.pdf